CLINICAL TRIAL: NCT02997722
Title: Ketamine: Its Effects on Suicidal Ideations and Inpatient Hospital Length of Stay
Brief Title: The Effect of Ketamine on the Length of Hospital Stay of Patients Hospitalized With Suicidal Ideation.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Staffing and space deficiencies prevented completion of the study.
Sponsor: Allen Richert (Other)
Responsible Party: Sponsor-Investigator, Allen Richert, Associate Professor of Psychiatry and Human Behavior, University of Mississippi Medical Center
Organization: University of Mississippi Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-0107
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Suicidal Ideation
Keywords: ketamine; suicidal ideation; length of stay
MeSH Terms: conditions — Suicidal Ideation | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine infusion (Experimental): Assignment to this arm involves receiving a single IV infusion of ketamine 0.5 mg/kg given over 45 minutes.
  Interventions: Drug: Ketamine
- Normal Saline infusion (Placebo Comparator): Assignment to this arm involves receiving an IV infusion of normal saline over the course of 45 minutes.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — IV infusion of ketamine 0.5 mg/kg administered over 45 minutes.
  Arms: Ketamine infusion
Drug: Normal Saline — IV infusion of 100 ml of normal saline over 45 minutes.
  Arms: Normal Saline infusion

SUMMARY:
This study will evaluate the effect of ketamine on the treatment of patients hospitalized with suicidal thoughts. Half of the patients will receive one dose of ketamine in the vein. The other half will receive a placebo. Because we think that ketamine will improve depression and suicidal thoughts, we expect that patients who receive ketamine will require less time in the hospital than patients who receive placebo.

DETAILED DESCRIPTION:
Patients admitted to UMMC's psychiatry inpatient unit with suicidal thoughts will be given the opportunity to participate in the study. Those patients who consent to participate, after being informed about the study and its risks, will be randomized to receive an IV infusion of either saline or ketamine 0.5 mg/kg. The infusion will be given within 24 hours of arriving on the psychiatry inpatient unit. We will record the dates and times that the patient was admitted to and discharged from the psychiatric inpatient unit. At completion of the study, we will compare the average length of stay, defined as date and time of discharge minus date of time of admission, of the group that received ketamine to the average length of stay of the group that received placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 64
2. Patients admitted to the University of Mississippi Medical Center inpatient psychiatry service with suicidal ideations

Exclusion Criteria:

1. Lifetime history of schizophrenia or other primary psychotic disorder
2. Current psychotic or manic symptoms
3. Substance use disorder within one month of admission
4. Positive urine toxicology at admission
5. Any lifetime abuse of ketamine or phencyclidine
6. Systolic BP >180 mmHg or diastolic BP >110 mmHg
7. Any patient who has eaten food within 8 hours prior to receiving the ketamine infusion or who has drank clear liquids within 2 hours prior to receiving the infusion
8. Known central nervous system (CNS) mass
9. CNS abnormalities
10. Hydrocephalus
11. Glaucoma
12. Acute globe injury
13. Porphyria
14. Untreated thyroid disease
15. Known coronary artery disease with poor functional capacity
16. Pregnancy
17. Currently breast-feeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen C Richert, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Infusion | Normal Saline Infusion
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Infusion | Normal Saline Infusion | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47.67 [38 to 59] | 36 [36 to 36] | 44.75 [36 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Inpatient Hospital Length of Stay
Description: We defined length of hospital stay as the difference between 1) the date and time that the patient was admitted to the psychiatry inpatient unit and 2) the date and time that the patient was discharged from the psychiatry inpatient.
Time Frame: The dates and times of each patients' admission to and discharge from the inpatient unit (i.e., the data necessary to calculate length of stay) were collected by chart review performed approximately 6 months after enrollment in the study.
Measure: Mean (Full Range); unit: hours
Arm/Group | Ketamine Infusion | Normal Saline Infusion
Number analyzed (Participants) | 3 | 1
hours | 130.75 [62.47 to 227.23] | 81.97 [81.97 to 81.97]

ADVERSE EVENTS:
Time Frame: We recorded adverse events that occurred during the infusion and for 30 minutes after the infusion.
Arm/Group | Ketamine Infusion | Normal Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Infusion (N=3) | Normal Saline Infusion (N=1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The small number of subjects (i.e., only 4) recruited prior to the premature termination of this study prevents one from drawing meaningful conclusions from this data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT02997722/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT02997722/Prot_SAP_001.pdf